CLINICAL TRIAL: NCT05567796
Title: Efficacy and Safety of Cagrilintide s.c. 2.4 Milligram (mg) in Combination With Semaglutide Subcutaneous (s.c). 2.4 mg (CagriSema s.c. 2.4 mg/2.4 mg) Once-weekly in Participants With Overweight or Obesity
Brief Title: A Research Study to See How Well CagriSema Helps People With Excess Body Weight Lose Weight
Acronym: REDEFINE 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4608; Universal Trial Number (UTN) (Other: U1111-1261-1912); 2020-005435-75 (EudraCT Number)
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cagrisema (Experimental): Participants will receive cagrilintide and semaglutide once-weekly after a dose escalation period of 16 weeks during the maintenance period for 52 weeks in the main phase. Participants randomised to this arm will be included in the extension phase for 97 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Cagrilintide (Active Comparator): Participants will receive cagrilintide s.c. and placebo matching to semaglutide once-weekly after a dose escalation period of 16 weeks during the maintenance period for 52 weeks.
  Interventions: Drug: Cagrilintide; Drug: Placebo semaglutide
- Semaglutide (Active Comparator): Participants will receive semaglutide s.c.and placebo matched to cagrilintide once-weekly after a dose escalation period of 16 weeks during the maintenance period for 52 weeks.
  Interventions: Drug: Semaglutide; Drug: Placebo cagrilintide
- Placebo s.c. (Placebo Comparator): Participants will receive placebo matched to cagrilintide and placebo matched to semaglutide once weekly for 68 weeks. Participants randomised to this arm will be included in the extension phase for 97 weeks.
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously.
  Arms: Cagrilintide; Cagrisema
Drug: Semaglutide — Participants will recieve semaglutide subcutaneously.
  Arms: Cagrisema; Semaglutide
Drug: Placebo cagrilintide — Participants will receive placebo matched to cagrilintide.
  Arms: Placebo s.c.; Semaglutide
Drug: Placebo semaglutide — Participants will receive placebo matched to semaglutide.
  Arms: Cagrilintide; Placebo s.c.

SUMMARY:
This study has 2 parts: First part is the main study and second part is the extension study. During the main study participants will receive 1 of 4 study medicines. If participants continue in the extension study, they will not receive any study medicine during the extension. The main study will look at how well CagriSema helps participants with excess body weight lose weight compared to a "dummy" medicine and 2 other medicines, cagrilintide and semaglutide. Participants will either get CagriSema, cagrilintide,semaglutide or "dummy" medicine. Which treatment participants get is decided by chance. They will take one injection once a week. The study medicine is injected briefly with a thin needle, typically in the stomach, thighs or upper arms.

Extension study: After the main study, not all participants will continue in the extension study. The study staff will tell the participant if they will continue or not into the extension study. In the extension study we will look at what happens to the participant's body weight and diseases related to excess body weight after the participant stops taking the study medicine. The main study will last for about 1½ years and the extension study will last for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age above or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) greater than or equal to 30.0 kilograms per square meter (kg/m^2) or b) BMI greater than or equal to 27.0 kg/m^2 with the presence of at least one weight-related comorbidity including, but not limited to hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease

Exclusion Criteria:

- Glycaemia related: a) Glycated Haemoglobin (HbA1c) greater than or equal to 6.5 percent (48 millimoles per mole [mmol/mol]) as measured by the central laboratory at screening b) History of type 1 or type 2 diabetes mellitus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
CagriSema versus placebo: Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
CagriSema versus placebo: Achievement of greater than or equal to (>=) 5% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants

SECONDARY OUTCOMES:
CagriSema versus placebo: Achievement of >= 20% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant
CagriSema versus placebo: Achievement of >= 25% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant
CagriSema versus placebo: Achievement of >= 30% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant
CagriSema versus cagrilintide and CagriSema versus semaglutide: Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage (%)
CagriSema versus placebo: Relative change in body weight | From baseline (week 0) to week 8
  Measured as percentage (%)
CagriSema versus placebo: Relative change in body weight | From baseline (week 0) to week 20
  Measured as percentage (%)
CagriSema versus placebo: Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeters (cm)
CagriSema versus placebo: Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeters of mercury (mmHg)
CagriSema versus placebo: Change in Impact of Weight on Quality Of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score.
CagriSema versus placebo: Change in SF-v2 Health Survey Acute (SF-36 v2 Acute) Physical Functioning Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. The SF-36v2 Acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2. Acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being.
CagriSema versus placebo, semaglutide and cagrilintide: Change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in kilograms (kg)
CagriSema versus placebo, semalutide and cagrilintide: Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilogram per square meter (kg/m^2)
CagriSema versus placebo, semaglutide and cagrilintide: Improvement in weight category | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants. The categories are: BMI, underweight less than (<) 18.5, normal weight 18.5 to <25, overweight 25.0 to <30, obesity class I 30 to < 35, obesity class II 35 to < 40, obesity class III >40.
CagriSema versus placebo: Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage (%)
CagriSema versus placebo: Change in HbA1c | From baseline (week 0) to end of treatment (week 68)
  Measured as millimoles per mole (mmol/mol).
CagriSema versus placebo: Change in Fasting Plasma Glucose (FPG) (mmol/L). | From baseline (week 0) to end of treatment (week 68)
  Measured as millimoles per liter (mmol/L).
CagriSema versus placebo: Change in FPG (mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured as milligrams per deciliter (mg/dL).
CagriSema versus placebo: Ratio to baseline in fasting serum insulin | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in mmHg
CagriSema versus placebo: Ratio to baseline in total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Ratio to baseline in High-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Ratio to baseline in Low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Ratio to baseline in Very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Ratio to baseline in Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Ratio to baseline in Free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus semaglutide and cagrilintide: Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeters (cm)
CagriSema versus semaglutide and cagrilintide: Change in SBP | From baseline (week 0) to end of treatment (week 68)
  Measured in mmHg
CagriSema versus semaglutide and cagrilintide: Ratio to baseline in total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus semaglutide and cagrilintide: Ratio to baseline in HDL | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus semaglutide and cagrilintide: Ratio to baseline in LDL | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus semaglutide and cagrilintide: Ratio to baseline in VLDL | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus semaglutide and cagrilintide: Ratio to baseline in Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus semaglutide and cagrilintide: Ratio to baseline in Free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
CagriSema versus placebo: Relative change in body weight (Measured in kilograms (kg)) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilograms (kg).
CagriSema versus placebo: Relative change in body weight (Measured in percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%).
CagriSema versus placebo: Absolute change in body weight (Measured in kilograms (kg)) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilograms (kg).
CagriSema versus placebo: Absolute change in body weight (Measured in percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%).
CagriSema versus placebo: Change in total fat mass by Dual energy X-ray absorption (DXA)a absolute to total body mass (Measured as kilograms (kg)) | From baseline (week 0) to end of treatment (week 68)
  Measured as kilograms (kg)
CagriSema versus placebo: Change in total fat mass by Dual energy X-ray absorption (DXA)a absolute to total body mass (Measured as percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage (%)
CagriSema versus placebo: Change in total fat mass by Dual energy X-ray absorption (DXA)a relative to total body mass (Measured as kilograms (kg)) | From baseline (week 0) to end of treatment (week 68)
  Measured as kilograms (kg)
CagriSema versus placebo: Change in total fat mass by Dual energy X-ray absorption (DXA)a relative to total body mass (Measured as percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage (%)
CagriSema versus placebo: Change in visceral fat mass by DXA, relative to baseline of fat mass in visceral fat mass region (Measured as percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage (%)
CagriSema versus placebo: Change in visceral fat mass by DXA, relative to baseline of fat mass in visceral fat mass region (Measured as %-points) | From baseline (week 0) to end of treatment (week 68)
  Measured as %-points
CagriSema versus placebo: Change in visceral fat mass by DXA, relative to total amount of fat mass in visceral fat mass region (Measured as percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage (%).
CagriSema versus placebo: Change in visceral fat mass by DXA, relative to total amount of fat mass in visceral fat mass region (Measured as %-points) | From baseline (week 0) to end of treatment (week 68)
  Measured as %-points
CagriSema versus placebo: Change in lean body mass by DXA absolute to total body mass (Measured in kilograms (kg)) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilograms (kg)
CagriSema versus placebo: Change in lean body mass by DXA absolute to total body mass (Measured in percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
CagriSema versus placebo: Change in lean body mass by DXA relative to total body mass (Measured in kilograms (kg)) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilograms (kg)
CagriSema versus placebo: Change in lean body mass by DXA relative to total body mass (Measured in percentage (%)) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
CagriSema versus placebo: Achievement of at least 14.6- point increase (yes/no) in IWQOL-Lite-CT Physical Function score | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score.
CagriSema versus placebo: Achievement of at least 3.7-point increase (yes/no) in SF-36v2 Physical Functioning score | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants. The SF-36v2 Acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2. Acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being.
CagriSema versus placebo: Change in IWQOL-Lite-CT - Physical Function Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score.
CagriSema versus placebo: Change in IWQOL-Lite-CT - Psychosocial Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score.
CagriSema versus placebo: Change in IWQOL-Lite-CT - Total Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score.
Change in Control of Eating (COEQ): Craving Control Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10).
Change in COEQ: Craving for Savoury food score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10).
Change in COEQ: Hunger score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10).
Change in COEQ: Craving for Sweets Score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10).
Change in COEQ: Positive Mood score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10).
Change in COEQ: Satiety score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. CoEQ is a 19-item multidimensional patient-reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10).
CagriSema versus placebo for subgroup with baseline PGI-S assessment 'Poor' : Change in IWQOL-Lite-CT Physical Function score | From baseline (week 0) to end of treatment (week 68)
  Measured as score points. IWQOL-Lite-CT version 3 is a 20-item COA instrument used to assess the impact of body weight changes in obesity studies on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score.
CagriSema versus placebo for subgroup with baseline PGI-S assessment 'Poor' : Achievement of at least 14.6-point increase (yes/no) in IWQOL-Lite-CT Physical Function score | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants.
CagriSema versus placebo, semalutide and cagrilintide: Ratio to baseline C-reactive protein (CRP) | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study-main part (week 75)
  Measured as count of events
Number of Treatment Emergent Serious adverse events (TESAEs) | From baseline (week 0) to end of study-main part (week 75)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (249):
- United States (44):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Velocity Clin Res Wstlke, Los Angeles, California
  - Univ of Colorado at Denver, Aurora, Colorado
  - New West Physicians,Inc., Golden, Colorado
  - Northeast Research Institute, Fleming Island, Florida
  - South Broward Research LLC, Miramar, Florida
  - Clinical Neuroscience Solution, Orlando, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Endeavor Health, Skokie, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Velocity Clinical Research Binghamton, Binghamton, New York
  - Comprehensive Weight Ctrl Prog, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Medication Mgmnt, LLC_Grnsboro, Greensboro, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare_NC, Raleigh, North Carolina
  - Accellacare, Wilmington, North Carolina
  - New Venture Medical Research, Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - The University of Penn Center, Philadelphia, Pennsylvania
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Medical Uni of SC Charleston, Charleston, South Carolina
  - Coastal Carolina Res Ctr, North Charleston, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group_Bristol, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Baylr Sctt White Rs Inst, Endo, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Health Res of Hampton Roads, Newport News, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
  - Rainier Clin Res Ctr Inc, Renton, Washington
- Argentina (6):
  - Fundación CESIM, Santa Rosa, La Pampa Province
  - CEDIC Centro de Investigación Clínica, CABA
  - Centro de Investigación Clínica, CABA
  - Centro Médico Viamonte SRL, CABA
  - Instituto Centenario, Ciudad de Buenos Aires
  - Sanatorio Norte, Santiago del Estero
- Australia (4):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Novatrials, Charlestown, New South Wales
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Momentum Clinical Research, Taringa, Queensland
- Belgium (8):
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - CHR Mons-Hainaut - Site Warquignies, Boussu
  - Cliniques Universitaires Saint-Luc - Serv Endocrinologie - Diabétologie, Brussels
  - UZ Antwerpen - UZA - Department of Endocrinology, Edegem
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Gent - Endocrinologie, Ghent
  - UZ Leuven - Endocrinology, Leuven
  - CHU Helora - Hôpital de Mons - Site Constantinople, Mons
- Bulgaria (16):
  - Medical centre Asclepius OOD, Dupnitsa, Kyustendil
  - "Multiprofile hospital for active treatment Puls" AD, Blagoevgrad
  - OCIPSOMC - Endocrinology NT EOOD, Montana
  - OCSOMCE - Dr. Albena Dinkova EOOD, Pleven
  - DCC Iztok EOOD, Plovdiv
  - ASOMCEM - Individual Practice - Dr. Antoanela Slavcheva, Rousse
  - ASOMCEM - IP - Dr. Antoanela Slavcheva, Rousse
  - Nader Yabrudi - ASMPVBE Individual practice, Smolyan
  - UMHAT "Aleksandrovska", Sofia
  - USHATE "Acad. Ivan Penchev" First Clinic of Endocrinology, Sofia
  - USHATE "Akad. Ivan Penchev" Second Clinic of Endocrinology, Sofia
  - DCC XVIII - Sofia EOOD, Sofia
  - "UMHAT "Tsaritsa Yoanna-ISUL"" EAD, Clinic of endocrinology and metabolic disease for metabolic disorders treatment, Sofia
  - "DCC XX - Sofia" EOOD, Endocrinology Consulting Room, Sofia
  - AIPSMC Dr. Artin Magardichyan EOOD, Varna
  - Medical center Berbatov, Yambol
- Canada (7):
  - C-endo Diab & Endo Clinic, Edmonton, Alberta
  - Synergy Wellness Clinic, Sherwood Park, Alberta
  - Ocean West Research Clinic, Surrey, British Columbia
  - Dr. M.B. Jones Inc, Victoria, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
- Denmark (7):
  - Aarhus Universitetshospital Diabetes og Hormonsygdomme, Aarhus N
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Center for Klinisk Metabolisk Forskning, Hellerup
  - Gentofte Hospital - Center for Klinisk Metabolisk Forskning, Hellerup
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
  - Sjællands Universitetshospital, Køge - Medicinsk Afdeling, Køge
  - Sjællands Universitetshospital, Køge
- Finland (4):
  - HUS Clinical Research Biomedicum 2U, Helsinki
  - Health Step Finland Oy, Kuopio
  - OYS - Sisätautien tutkimusyksikkö, Oulu
  - Turku University Hospital, Turku
- France (5):
  - Aphp-Hopital La Pitie Salpetriere-3, Paris
  - Hospices Civils de Lyon-Hopital Lyon Sud-1, Pierre-Bénite
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Les Hopitaux Universitaires de Strasbourg-Hopital de Hautepierre-1, Strasbourg
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (9):
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Uniklinik Leipzig - Klinik und Poliklinik für Endokrinologie, Nephrologie, Rheumatologie, Leipzig
  - AmBeNet GmbH, Leipzig
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - MZM Praxis Drs. Erlinger, Stuttgart
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- India (19):
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Sir H. N. Reliance Foundation Hospital and Research Centre, Mumbai, Maharashtra
  - Wockhardt Hospital, Mumbai Central, Mumbai, Maharashtra
  - Government Medical College and Super Speciality Hospital, Nagpur, Nagpur, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - chelleram Diabetes Institute, Pune, Maharashtra
  - Maulana Azad Medical College, Delhi, New Delhi
  - Post Graduate Institute of Medical Education & Research_Chandigarh, Chandigarh, Punjab
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Eternal Heart Care Centre, Jaipur, Rajasthan
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - AIG Hospitals,Hyderabad, Hyderabad, Telangana
  - All India Institute of Medical Sciences_New Dehli, Delhi
  - Osmania General Hospital, Hyderabad
- Italy (11):
  - A.O.U. Consorziale Policlinico di Bari, Bari, BA
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - Policlinico San Donato S.p.A., San Donato Milanese (MI), Lombardy
  - Pol. Uni. Campus Biomedico, Roma, RM
  - Azienda Ospedaliera Universitaria Senese, Siena, SI
  - A.O.Universitaria S.ORSOLA-MALPIGHI - U.O.Endocrinologia e Cura, Bologna
  - ARNAS Garibaldi Catania - Presidio Ospedaliero Garibaldi-Centro, Catania
  - Azienda Ospedaliera di Padova Clin.Med.3, Padua
  - Ospedale Civico Partinico di Palermo, Partinico
  - Policlinico Universitario Tor Vergata, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Roma
- Japan (15):
  - Shinsapporo Seiryou Hospital_General Clinical Department, Sapporo, Hokkaido
  - OCROM Clinic_Internal medicine, Suita-shi, Osaka
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Chiba University Hospital_Diabetes, Metabolism and Endocrinology, Chiba-shi, Chiba
  - Kawada Clinic, Gunma
  - Motomachi Takatsuka Naika Clinic_Internal Medicine, Kanagawa
  - Osaka NISHI-UMEDA Clinic_Internal Medicine, Osaka
  - Asano Clinic, Saitama
  - Shinden Higashi Clinic, Sendai-shi, Miyagi
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Miho Clinic, Tokyo
  - ToCROM Clinic_Internal Medicine, Tokyo
  - Higashi-shinjuku clinic, Tokyo
- Mexico (5):
  - Consultorio Arechavaleta Granell María del Rosario, Guadalajara, Jalisco
  - Centro de Investigacion Clinica Endocrinologica de Jalisco, Guadalajara, Jalisco
  - Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Cardiolink Clin Trials S.C., Monterrey, Nuevo León
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Spaarne Gasthuis_Hoofddorp, Hoofddorp
  - Bravis Ziekenhuis, Roosendaal
  - Albert Schweitzer Ziekenhuis, locatie Zwijndrecht, Zwijndrecht
- Poland (21):
  - 50BIO.COM Sp. z o.o., Bydgoszcz, Kujawsko-Pomorskie Voivodeship
  - Gierach-Med, Bygdoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Beata Miklaszewicz & Dariusz Dabrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - Terpa Sp. z o.o. Sp. k., Lublin, Lubelskie Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Im. Prof. W. Orłowskiego Centrum Medycznego Kształcenia Podyplomowego, Warsaw, Masovian Voivodeship
  - Instytut Diabetologii Sp. z o.o., Warsaw, Mazovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok, Podlaskie Voivodeship
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Salvia, Katowice, Slaskie Voivodeship
  - Klinika Bellamed, Elblag, Warmian-Masurian Voivodeship
  - Centrum Ginekologii, Poloznictwa i Leczenia Nieplodnosci, Poznan, Wielkopolskie Voivodeship
  - Centrum Ginekologii, Położnictwa i Leczenia Niepłodności, Poznan, Wielkopolskie Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship
  - Centrum Medyczne Plejady, Krakow
  - Beata Mikłaszewicz & Dariusz Dąbrowski "CARDIAMED" s.j., Legnica
  - Terpa Sp. z o.o. Sp. k., Lublin
  - Samodzielny Publiczny Szpital Kliniczny Im. Prof. W. Orłowskiego Centrum Medycznego Kształcenia Podyplomowego, Warsaw
  - Instytut Diabetologii Sp. z o.o., Warsaw
- Serbia (4):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad
- South Africa (9):
  - East Rand Physicians, Benoni, Gauteng
  - Dr R Dulabh, Johannesburg, Gauteng
  - Dr Moosa's Rooms, Lenasia, Gauteng
  - Shop#1 Health Emporium, Midrand, Gauteng
  - Botho ke Bontle Health Services, Pretoria, Gauteng
  - Dr Vawda's site, Durban, KwaZulu-Natal
  - Dr J Reddy, Durban, KwaZulu-Natal
  - Armansis Medical Centre, Brits, North West
  - Dr Hilton Kaplan, Cape Town, Western Cape
- South Korea (11):
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - The catholic university of Korea, Bucheon St.Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (7):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de León, León
  - Hospital Gregorio Marañón, Madrid
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Infanta Luisa, Seville
  - Hospital Vithas Sevilla, Seville
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital_main, Taipei
- Turkey (Türkiye) (16):
  - Baskent University Ankara Hospital, Ankara, Cankaya
  - Başkent Üniversitesi Ankara Hastanesi-Aile Hekimliği, Ankara, Cankaya
  - Haseki Egitim ve Arastirma Hastanesi, Sultangazi, Istanbul
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Adana
  - Başkent Üniversitesi Adana Dr. Turgut Noyan Uygulama ve Araştırma Merkezi, Adana
  - Ankara Bilkent Şehir Hastanesi-Dahiliye, Ankara
  - Ankara Sehir Hastanesi Dahiliye Klinigi, Ankara
  - Akdeniz Üniversitesi Hastanesi- Endokrinoloji, Antalya
  - Hatay Mustafa Kemal Universitesi Saglik Uygulama ve Arastirm, Hatay
  - Istanbul Universitesi Istanbul Tip Fakultesi - Endokrinoloji, Istanbul
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Endokrinoloji, Istanbul
  - Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi- Endokrinoloji, Istanbul
  - Haydarpaşa Numune Eğitim ve Araştırma Hastanesi - Endokrinoloji, Istanbul
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - Sivas Cumhuriyet Univesity Endocrinology Department, Sivas
  - Sivas Cumhuriyet Üniversitesi Hastanesi -Endokrinoloji, Sivas
- United Kingdom (14):
  - Princess Royal University Hospital, Orpington, Kent
  - Layton Medical Centre, Blackpool
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - Countess of Chester Hospital, Chester
  - Hathaway Medical Centre, Chippenham
  - University Hospital Coventry - WISDEM Centre, Coventry
  - Aintree University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - Guys Hospital, London
  - Imperial College London, London
  - UCL - Obesity, London
  - Princess Royal University Hospital, Orpington
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Verma S, Bottcher M, Brown P, Dicker D, Rubino D, Sbraccia P, Sharma AM, Smedegaard L, Sorrig R, Garvey WT. CagriSema Reduces Blood Pressure in Adults With Overweight or Obesity: REDEFINE 1. Hypertension. 2026 Feb;83(2):e26055. doi: 10.1161/HYPERTENSIONAHA.125.26055. Epub 2025 Dec 2. PMID 41328546
- [Derived] Garvey WT, Bluher M, Osorto Contreras CK, Davies MJ, Winning Lehmann E, Pietilainen KH, Rubino D, Sbraccia P, Wadden T, Zeuthen N, Wilding JPH; REDEFINE 1 Study Group. Coadministered Cagrilintide and Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2025 Aug 14;393(7):635-647. doi: 10.1056/NEJMoa2502081. Epub 2025 Jun 22. PMID 40544433